CLINICAL TRIAL: NCT01610570
Title: Phase I/II Trial of Mithramycin in Children and Adults With Refractory Extracranial Solid Tumors (Phase I) or Ewing Sarcoma and EWSFLI1 Fusion Transcript (Phase II)
Brief Title: Mithramycin for Children and Adults With Solid Tumors or Ewing Sarcoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was closed to enrollment before dose level one was completed.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brigitte Widemann, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120135; 12-C-0135
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2017-12

CONDITIONS: Ewing Sarcoma; Sarcoma
Keywords: Dose Limiting Toxicity; Maximum Tolerated Dose; Radiographic Response; Time to Progression; Bone Tumors
MeSH Terms: conditions — Sarcoma, Ewing; Sarcoma; Bone Neoplasms | interventions — Plicamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I Dose Level -1 (Experimental): Dose Escalation Phase 9.0 mcg/kg.dose
  Interventions: Drug: Mithramycin
- Phase I Dose Level 1 (Experimental): Dose Escalation Phase 13.0 mcg/kg.dose
  Interventions: Drug: Mithramycin
- Phase I Dose Level 2 (Experimental): Dose Escalation Phase 17.5 mcg/kg.dose
  Interventions: Drug: Mithramycin
- Phase II - Expansion Phase (Experimental): Expansion phase 17.5 mcg/kg.dose
  Interventions: Drug: Mithramycin

INTERVENTIONS:
Drug: Mithramycin — Phase I Portion: Mithramycin will be administered in escalating doses to children and adolescents intravenously over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Phase differs from the recommended adult dose for Phase II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously. Phase II Portion: mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults.

SUMMARY:
Background:

- Mithramycin is a drug that was first tested as a cancer therapy in the 1960s. It acted against some forms of cancer, but was never accepted as a treatment. Research suggests that it may be useful against some solid tumors, particularly Ewing sarcoma. Researchers want to see if mithramycin can be used to treat solid tumors in children and adults. It will be tested in different groups of people, including those with a type of Ewing sarcoma that contains a chemical called Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1).

Objectives:

- To see if mithramycin is safe and effective against solid tumors and Ewing sarcoma in children and adults.

Eligibility:

* Children and young adults between 1 and 17 years of age with solid tumors that have not responded to standard treatment.
* Adults at least 18 years of age with EWS-FLI1 Ewing sarcoma that has not responded to standard treatment.
* Children and young adults between 1 and 17 years of age with EWS-FLI1 Ewing sarcoma that has not responded to standard treatment.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies and tumor tissue samples will be used to monitor the cancer before treatment. Individuals with solid brain tumors will not be eligible.
* Participants will receive mithramycin every day for 7 days, followed by 14 days without treatment. Each 28-day round of treatment is called a cycle.
* Treatment will be monitored with frequent blood tests and imaging studies.
* Participants will continue to take the drug for as long as the side effects are not severe and the tumor responds to treatment.

DETAILED DESCRIPTION:
BACKGROUND:

* Mithramycin, an anti-tumor antibiotic, underwent broad clinical evaluation in solid tumors and leukemias in the 1960s and demonstrated activity in some leukemias, lymphomas, and solid tumors. In particular, mithramycin was found to have activity against testicular cancers and was briefly used in the clinic for this tumor prior to the development of the currently used treatment regimen.
* The Ewing Sarcoma Family of Tumors (ESFT) is the second most common malignant bone tumor of childhood. There has been very little improvement in overall patient survival in past years, particularly for patients with high risk metastatic or relapsed disease. Therefore, there is a need for effective novel agents for the treatment of this disease.
* Multiple studies have shown that suppressing the expression of EWS-FLI1 effectively limits the tumorigenicity of ESFT cells. Laboratory studies have shown that mithramycin effectively suppresses the activity of EWS-FLI1 both in vitro and in vivo.

OBJECTIVES (PRIMARY):

* Phase I portion of this study is to: determine the tolerability, toxicity, and the recommended phase II dose of mithramycin in children and adolescents with refractory extracranial solid tumors.
* Phase II portion of this trial is to: determine the objective response rate (complete response (CR) and partial response (PR)) of Ewing sarcoma to mithramycin in children and adults using Response Evaluation Criteria in Solid Tumors (RECIST) criteria when administered at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression.
* Phase II portion of this trial to: evaluate if mithramycin inhibits NR0B1 in tumor tissue and determine changes in gene expression signature pre-treatment and at steady state on day +4 of treatment in patients greater than or equal to 18 years old with Ewing sarcoma and EWS/FLI1 fusion transcript with disease amenable to percutaneous biopsy.

ELIGIBILITY:

* Phase I Portion: children (greater than or equal to 12 months) and adolescents (less than or equal to 17 years) with recurrent or refractory extracranial solid tumors.
* Phase II Portion in adults: adults (greater than or equal to 18 years of age at enrollment) with recurrent or refractory measurable extracranial Ewing sarcoma and the EWS-FLI1 fusion transcript.
* Phase II Portion in children and adolescents: Once the adult dose is deemed safe, children

(greater than or equal to 12 months) and adolescents (less than or equal to 17 years) with recurrent or refractory measurable

extracranial Ewing sarcoma and the EWS-FLI1 fusion transcript will begin enrollment to the Phase II portion.

* Participants must meet safety laboratory criteria and prior therapy limitations.

DESIGN:

Phase I Portion: Mithramycin will be administered in escalating doses to children and adolescents intravenously over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. The cohort at the recommended dose or maximum tolerated dose (MTD) will be expanded up to 12 patients, and attempts will be made to enroll 6 patients that are greater than or equal to 12 years of age and 6 patients that are < 12 years of age to gain experience with a broad age range of patients. A maximum of 18 evaluable patients will be enrolled on the phase I portion.

* Phase II Portion: Using a Simon two stage design, mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every

  28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with EWS-FLI1 fusion transcript. Up to 24 evaluable patients will be enrolled on the phase II portion.
* The Phase I and Phase II portions of the protocol will enroll patients simultaneously.

ELIGIBILITY:
* INCLUSION CRITERIA
* Diagnosis
* Patients current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
* Phase I Portion: Measurable or evaluable refractory or recurrent extracranial solid tumors, excluding brain tumors and cerebral metastases.
* Phase II Portion adults and children: Refractory or recurrent extracranial Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript. Patients enrolled to this cohort must have measurable disease. Presence of the transcript will be determined during histologic confirmation of disease with a Clinical Laboratory Improvement Amendments (CLIA) approved EWS-FLI paraffin assay in the Laboratory of Pathology Center for Cancer Research, National Cancer Institute (CCR, NCI), unless a pathology report documenting presence of the transcript using a CLIA approved assay is obtained from the referring institution.
* Histologic confirmation of disease in the Laboratory of Pathology, CCR, NCI, National Institutes of Health (NIH).
* Age
* Phase I Portion: greater than or equal to 12 months to less than or equal to 17 years
* Phase II Portion in adults initially: greater than or equal to 18 years
* Phase II Portion expanded in pediatrics after determination of phase II dose in children will include children greater than or equal to 12 months to less than or equal to 17 years
* Performance Score: Karnofsky (> 10-17 years old) or Lansky (less than or equal to 10 years old) greater than or equal to 50%, or Eastern Cooperative Oncology Group (ECOG) 1 or 2 (adults)
* Prior therapy
* greater than or equal to 2 weeks must have elapsed since local palliative radiation (XRT) (small port);
* greater than or equal to 24 weeks must have elapsed since prior total body irradiation (TBI), craniospinal XRT, or if greater than or equal to 50%
* radiation of pelvis;
* greater than or equal to 6 weeks must have elapsed since other substantial BM radiation;
* greater than or equal to 12 weeks must have elapsed since stem cell transplant or infusion without TBI and no active graft vs. host disease;
* greater than or equal to 3 weeks must have elapsed from last dose of myelosuppressive chemotherapy (six

weeks for nitrosoureas);

at least 3 half-lives must have elapsed since monoclonal antibody1;(https://members.childrensoncologygroup.org/Disc/devtherapeutics/default.asp for listing of monoclonal antibody half-lives.)

* greater than or equal to 7 days must have elapsed from the last dose of biologic agents.
* greater than or equal to 7 days since the completion of therapy with a growth factor
* Recovered from acute toxicities of prior therapy to less than or equal to Grade 1; specifically

  a) Hematologic and Coagulation Parameters

  i. Peripheral absolute neutrophil count (ANC) greater than or equal to 1000/mcL

ii. Platelets greater than or equal to 75,000/ mcL (transfusion independent)

iii. Hemoglobin greater than or equal to 8 g/dL (packed red blood cell (PRBC) transfusions permitted)

iv. Normal prothrombin time (PT)/partial thromboplastin time (PTT) with the exception of a lupus anticoagulant, which is permitted, may be corrected with Vitamin K administration or transfusion. Fibrinogen greater than or equal to the lower limit of normal.

b) Hepatic Function

i. Bilirubin (total) less than or equal to 1.5 times upper limit of normal (ULN)

ii. Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase (SGPT) less than or equal to 3.0 times ULN

iii. Albumin > 2 g/dL

c) Renal Function

i. Creatinine clearance greater than or equal to 60 mL/min/1.73 m^2, or serum creatinine base on age and gender as follows:

Age (years) Maximum Serum Creatinine (mg/dL)

2 to < 6 0.8 0.8

6 to < 10 1 1

10 to < 13 1.2 1.2

13 to < 16 1.5 1.4

greater than or equal to 16 1.7 1.4

* Normal calcium, magnesium and phosphorus (can be on oral supplementation
* Cardiac Function: Left ventricular ejection fraction (EF) within normal institutional limits by Echocardiogram or multi-gated acquisition scan (MUGA)
* Ability to give informed consent. For patients < 18 years of age their legal guardian must give informed consent. Pediatric patients will be included in age appropriate discussion in order to obtain verbal assent.
* Female and male patients (and when relevant their partners) must be willing to practice birth control (including abstinence) during and for two months after treatment, if of childbearing potential during sexual contact with a female of childbearing potential.
* A durable power of attorney (DPA) will be offered to all patients greater than or equal to 18 years old.
* Eligibility criteria for mandatory serial tumor biopsies
* Age: greater than or equal to 18 years old
* Ewing sarcoma with EWS-FLI1 fusion transcript
* Hematologic and coagulation parameters within 2 days prior to each biopsy: Normal PT/PTT with exception of lupus anticoagulant, platelets greater than or equal to 75,000/mcL, peripheral ANC greater than or equal to 750/mcL
* Willing to undergo biopsies, which will only be performed on tumors amenable to percutaneous biopsy

EXCLUSION CRITERIA:

* Clinically significant systemic illness (e.g. serious active infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the judgment of the PI would compromise the patient s ability to tolerate protocol therapy or significantly increase the risk of complications.
* Patients with a history intracranial Ewing sarcoma including cerebral metastases
* Patients with evidence of active bleeding, intratumoral hemorrhage or history of bleeding diatheses
* Patients who are receiving anticoagulants other than prophylactic anticoagulation of venous or arterial access devices, provided that requirements for PT, PTT and fibrinogen are met, as described
* Investigational Drugs: Patients who are currently receiving another investigational drug
* Patients who are concurrently receiving agents, which may increase the risk for mithramycin related toxicities, such as hemorrhage including:
* Thrombolytic agents
* Anti-inflammatory drugs, nonsteroidal (nonsteroidal anti-inflammatory drugs (NSAIDs)) or aspirin or salicylate containing products, which may increase risk of hemorrhage
* Dextran
* Dipyridamole
* Sulfinpyrazone
* Valproic acid
* Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents
* Lactating or pregnant females (due to risk to fetus or newborn, and lack of testing for excretion in breast milk).
* Patients with history of human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) due to potentially increased risk of mithramycin toxicity in this population.
* Hypersensitivity to plicamycin (mithramycin)
* Requirement for any of the contraindicated medications: nonsteroidal anti-inflammatory drugs, aspirin, dextran or other iron containing solutions (due to incompatibility), dipyridamole, sulfinpyrazone or valproic acid
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Patients receiving concurrently other therapies directed at their cancer.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-05-10 (Actual); Primary Completion 2014-05-21 (Actual); Study Completion 2014-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esiashvili N, Goodman M, Marcus RB Jr. Changes in incidence and survival of Ewing sarcoma patients over the past 3 decades: Surveillance Epidemiology and End Results data. J Pediatr Hematol Oncol. 2008 Jun;30(6):425-30. doi: 10.1097/MPH.0b013e31816e22f3. PMID 18525458
- [Background] Delattre O, Zucman J, Melot T, Garau XS, Zucker JM, Lenoir GM, Ambros PF, Sheer D, Turc-Carel C, Triche TJ, et al. The Ewing family of tumors--a subgroup of small-round-cell tumors defined by specific chimeric transcripts. N Engl J Med. 1994 Aug 4;331(5):294-9. doi: 10.1056/NEJM199408043310503. PMID 8022439
- [Background] Delattre O, Zucman J, Plougastel B, Desmaze C, Melot T, Peter M, Kovar H, Joubert I, de Jong P, Rouleau G, et al. Gene fusion with an ETS DNA-binding domain caused by chromosome translocation in human tumours. Nature. 1992 Sep 10;359(6391):162-5. doi: 10.1038/359162a0. PMID 1522903
- [Result] Grohar PJ, Glod J, Peer CJ, Sissung TM, Arnaldez FI, Long L, Figg WD, Whitcomb P, Helman LJ, Widemann BC. A phase I/II trial and pharmacokinetic study of mithramycin in children and adults with refractory Ewing sarcoma and EWS-FLI1 fusion transcript. Cancer Chemother Pharmacol. 2017 Sep;80(3):645-652. doi: 10.1007/s00280-017-3382-x. Epub 2017 Jul 22. PMID 28735378
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0135.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was closed to enrollment before dose level I was completed and hence no patients were enrolled on other dose levels.
Groups:
- Phase I Dose Level -1: Dose Escalation Phase
  9.0 mcg/kg/dose Phase I Portion: Mithramycin will be administered in escalating doses to children and adolescents intravenously over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Phase differs from the recommended adult dose for Phase II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously
- Phase 1 Dose Level 1: Dose Escalation Phase
  13.0 mcg/kg/dose Phase I Portion: Mithramycin will be administered in escalating doses to children and adolescents intravenously over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Phase differs from the recommended adult dose for Phase II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously
- Phase 1 Dose Level 2: Dose Escalation Phase
  17.5 mcg/kg/dose Phase I Portion: Mithramycin will be administered in escalating doses to children and adolescents intravenously over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Phase differs from the recommended adult dose for Phase II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously
- Phase II - Expansion Phase: Expansion phase 17.5 mcg/kg.dose Mithramycin: Phase I Portion: Mithramycin will be administered in escalating doses to children and adolescents intravenously over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Phase differs from the recommended adult dose for Phase II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously.
Period: Ph I >/= 12 mo. Children & Adolescents
Arm/Group | Phase I Dose Level -1 | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase II - Expansion Phase
Started | 0 | 2 | 0 | 0
Completed | 0 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Ph II >/= 18yrs of Age at Enrollment
Arm/Group | Phase I Dose Level -1 | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase II - Expansion Phase
Started | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Ph II >/= 12 mo. & </=17yrs
Arm/Group | Phase I Dose Level -1 | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase II - Expansion Phase
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I Dose Level 2: Dose Escalation Phase 17.5 mcg/kg/dose Phase I Portion: Mithramycin will be administered in escalating doses to children and adolescents intravenously over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Phase differs from the recommended adult dose for Phase II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously
- Phase 2: Expansion phase 17.5 mcg/kg.dose Mithramycin: Phase I Portion: Mithramycin will be administered in escalating doses to children and adolescents intravenously over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Phase differs from the recommended adult dose for Phase II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously.
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level -1 | Phase 1 Dose Level 1 | Phase I Dose Level 2 | Phase 2 | Total
Number analyzed (Participants) | 0 | 2 | 0 | 6 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 2 |  | 0 | 2
  Between 18 and 65 years |  | 0 |  | 6 | 6
  >=65 years |  | 0 |  | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 12.5 (0) |  | 23.8 (5.3) | 21.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 |  | 3 | 3
  Male |  | 2 |  | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 1 |  | 0 | 1
  Not Hispanic or Latino |  | 1 |  | 6 | 7
  Unknown or Not Reported |  | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 |  | 0 | 0
  Asian |  | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 |  | 0 | 0
  Black or African American |  | 0 |  | 0 | 0
  White |  | 2 |  | 6 | 8
  More than one race |  | 0 |  | 0 | 0
  Unknown or Not Reported |  | 0 |  | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 2 |  | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Mithramycin
Description: The MTD will be the maximum dose at which fewer than one-third of patients experience Dose Limiting Toxicity (DLT) (i.e., non-hematologic toxicity and hematologic toxicity) during cycle 1 (or 28 days) of therapy.
Time Frame: Cycle 1 of therapy (or 28 days)
Population: MTD was not determined because based on pharmacokinetic data, a clinically relevant dose could not be obtained with the dose strategy. A minimum of 3 patients must be enrolled on a dose level to complete that dose level. Because only 2 patients were enrolled on phase I portion of the trial, dose level 1 was not completed and an MTD was not reached.
Groups:
- Phase I Dose Level -1: Dose Escalation Ph 9.0 mcg/kg dose Ph I: Mithramycin will be administered in escalating doses to children and adolescents intravenously IV) over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Ph differs from the recommended adult dose for Ph II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered IV at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously. Ph II: mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults.
- Phase I Dose Level 1: Dose Escalation Phase 13.0 mcg/kg.dose Ph I: Mithramycin will be administered in escalating doses to children and adolescents intravenously IV) over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Ph differs from the recommended adult dose for Ph II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered IV at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously. Ph II: mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults.
- Phase I Dose Level 2: Dose Escalation Phase 17.5 mcg/kg.dose Ph I: Mithramycin will be administered in escalating doses to children and adolescents intravenously IV) over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Ph differs from the recommended adult dose for Ph II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered IV at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously. Ph II: mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults.
Arm/Group | Phase I Dose Level -1 | Phase I Dose Level 1 | Phase I Dose Level 2
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events. For a detailed list of serious and non-serious adverse events see the adverse event module.
Time Frame: 95 days
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Dose Level -1: Dose Escalation Phase 9.0 mcg/kg.dose Ph I: Mithramycin will be administered in escalating doses to children and adolescents intravenously IV) over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Ph differs from the recommended adult dose for Ph II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered IV at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously. Ph II: mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults.
- Phase II - Expansion Phase: Expansion phase 17.5 mcg/kg.dose Ph I: Mithramycin will be administered in escalating doses to children and adolescents intravenously IV) over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Ph differs from the recommended adult dose for Ph II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered IV at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously. Ph II: mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults.
Arm/Group | Phase I Dose Level -1 | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase II - Expansion Phase
Number analyzed (Participants) | 0 | 2 | 0 | 6
Participants |  | 2 |  | 6

3. Secondary Outcome: Objective Response Rate (Complete Response (CR) + Partial Response (PR))
Description: Objective response in children and adolescents with Ewings sarcoma - friend leukemia integration 1 transcription factor to mithramycin is defined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions.
Time Frame: 1-2 months
Population: This is a phase II objective, thus phase I groups are not shown here.
Measure: Number; unit: participants
Arm/Group | Phase II - Expansion Phase
Number analyzed (Participants) | 6
participants
  Complete response (CR) | 0
  Partial response (PR) | 0

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the number of days from enrollment until disease progression, death because of treatment complications, resection of measureable tumor, or last patient follow-up, whichever comes first, assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (Note: the appearance of one or more new lesions is also considered progressions). Stable disease (SD) is neither shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: At date of progression, an average of 56 days
Population: TTP was not evaluated for patients on the phase I portion of the study (patients 4 and 6). TTP was evaluated on the phase II portion of the study only for patients 1, 2, 3, 5, 7, and 8.
Measure: Number; unit: Days
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase II - Expansion Phase
Number analyzed (Participants) | 0 | 0 | 6
Days
  Patient #1 |  |  | 56
  Patient #2 |  |  | 56
  Patient #3 |  |  | 126
  Patient #5 |  |  | 54
  Patient #7 |  |  | 56
  Patient #8 |  |  | 56

5. Secondary Outcome: Count of Participants With NR0B1 Expression in Tumor Biopsies
Description: Biopsies were to be obtained in adult patients who have disease that could be safely biopsied.
Time Frame: Pre-treatment and day 4 (+/- 1 day)
Population: This outcome measure was not done because none of the adult patients on this study had disease that was deemed accessible.
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase II - Expansion Phase
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With a Change in Tumor Burden Measured by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Measurable disease were to be quantified using volumetric magnetic resonance imaging analysis per the RECIST, measuring soft tissue disease. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes. Complete response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (Note: the appearance of one or more new lesions is also considered progressions). Stable disease (SD) is neither shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: ≥4 weeks from baseline
Population: Changes in tumor burden was not evaluated for patients on the phase I portion of the study (patients 4 and 6). Changes in tumor burden was evaluated on the phase II portion of the study only for patients 1, 2, 3, 5, 7, and 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase II - Expansion Phase
Number analyzed (Participants) | 0 | 0 | 6
Participants
  Complete Response |  |  | 0
  Partial Response |  |  | 0
  Progressive Disease |  |  | 6
  Stable Disease |  |  | 0

7. Secondary Outcome: Number of Participants With a Change in Tumor Burden Measured by the World Health Organization (WHO) Criteria
Description: Per the WHO criteria, progressive disease is a 25% increase in tumor lesions, or the appearance of any new measureable or non-measureable tumor lesions. Partial response is ≥50% decrease in tumor lesions. Complete response is disappearance of all tumor lesions. Stable disease is 50% decrease in tumor lesions compared to baseline, nor 25% increase compared with nadir.
Time Frame: ≥4 weeks from baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase II - Expansion Phase
Number analyzed (Participants) | 0 | 0 | 6
Participants
  Complete Response |  |  | 0
  Partial Response |  |  | 0
  Progressive Disease |  |  | 6
  Stable Disease |  |  | 0

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Mithramycin Using Non-Compartmental Methods
Description: The maximum observed analyte concentration in serum was reported. Mithramycin plasma concentrations were measured using high-performance liquid chromatography tandem mass spectroscopic method, and analysis was performed using the Phoenix 6.3 with WinNonlin noncompartmental method.
Time Frame: Prior to dose 1, 3hrs after dose 1 infusion, prior to end of 6hr infusion, 0.25, 0.5, 1,2,3,4,5, & 7hr post infusion, & between 9 & 12hr completion of 1st dose infusion. Trough & end of infusion samples obtained w/day 2,4,&7 doses & 24hr after day 7 dose
Population: After dose-limiting hepatotoxicity was observed in the 1st 2 adult patients (pts), the protocol was subsequently amended to allow PK analysis prior to and at the completion of the first dose during cycle 1 on both the ph 1 & 2 portions of the trial in consenting pts. PK sampling was not mandatory, thus not all pts (i.e. 4/8 pts) had PK analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Phase I Dose Level 1 & Phase II Expansion Phase: Dose levels 13.0 and 17.5 mcg/kg. dose Ph I: Mithramycin will be administered in escalating doses to children and adolescents intravenously IV) over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression. If maximum tolerated dose (MTD) in this Ph differs from the recommended adult dose for Ph II, the protocol will be amended. Using a Simon two stage design, mithramycin will be administered IV at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults with Ewing sarcoma with Ewings sarcoma - friend leukemia integration 1 transcription factor (EWS-FLI1) fusion transcript Both Phases will enroll patients simultaneously. Ph II: mithramycin will be administered intravenously at 17.5 microgram/kg over 6 hours once daily for 7 days to be repeated every 28 days until unacceptable toxicity or disease progression to children and adults.
Arm/Group | Phase I Dose Level 1 & Phase II Expansion Phase
Number analyzed (Participants) | 4
ng/mL | 17.8 (4.6)

9. Secondary Outcome: Half-Life (HL) of Mithramycin
Description: Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half. Analysis was performed using the Phoenix 6.3 with WinNonlin noncompartmental method.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase I Dose Level 1 & Phase II Expansion Phase
Number analyzed (Participants) | 4
hours | 6.8 (2.3)

10. Secondary Outcome: Area Under the Curve Extrapolated to Infinity (AUCinf)
Description: AUC is a measure of the serum concentration of mithramycin over time. It is used to characterize drug absorption. Analysis was performed using the Phoenix 6.3 with WinNonlin noncompartmental method.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Phase I Dose Level 1 & Phase II Expansion Phase
Number analyzed (Participants) | 4
h*ng/mL | 1544 (754)

11. Secondary Outcome: Area Under the Curve for the Dosing Interval (AUCtau)
Description: AUCtau is AUC for the dosing interval. Analysis was performed using the Phoenix 6.3 with WinNonlin noncompartmental method.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Phase I Dose Level 1 & Phase II Expansion Phase
Number analyzed (Participants) | 4
h*ng/mL | 394 (94)

12. Secondary Outcome: Clearance at Steady State (CLss)
Description: The CL is a quantitative measure of the rate at which a drug substance is removed from the body. Analysis was performed using the Phoenix 6.3 with WinNonlin noncompartmental method.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Phase I Dose Level 1 & Phase II Expansion Phase
Number analyzed (Participants) | 4
L/h | 1.9 (0.8)

13. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Analysis was performed using the Phoenix 6.3 with WinNonlin noncompartmental method.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Phase I Dose Level 1 & Phase II Expansion Phase
Number analyzed (Participants) | 4
L | 293 (88)

14. Other Pre Specified Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: Hematologic DLT was defined as any grade 4 neutropenia (<500/µL) or thrombocytopenia (<25,000/µL) refractory to platelet transfusion, any grade 2 bleeding not promptly (within 6 h of appropriate intervention) corrected with blood product support. Non-hematologic DLT's were any mithramycin-related grade ≥3 toxicity with the exception of grade 3 nausea, vomiting, or diarrhea that was controlled by symptomatic treatment within 72h, asymptomatic grade 3 elevation of serum transaminases that return to ≤grade 1 within 14 days of completing mithramycin administration, and asymptomatic electrolyte abnormalities that are correctable to grade2 or less within 48h.
Time Frame: Cycle 1 of therapy (or 28 days)
Population: Hepatotoxicity
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase II - Expansion Phase
Number analyzed (Participants) | 2 | 0 | 6
Participants | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: 95 days
Arm/Group | Phase I Dose Level -1 | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase II - Expansion Phase
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2 | 0/0 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/2 | 0/0 | 1/6
Other Adverse Events (participants affected / at risk) | 0/0 | 2/2 | 0/0 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level -1 (N=0) | Phase I Dose Level 1 (N=2) | Phase I Dose Level 2 (N=0) | Phase II - Expansion Phase (N=6)
Fever (General disorders) | 0 | 0 | 0 | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 1 (1)
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level -1 (N=0) | Phase I Dose Level 1 (N=2) | Phase I Dose Level 2 (N=0) | Phase II - Expansion Phase (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 | 1 (4) | 0 | 6 (32)
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 (2)
Anemia (Blood and lymphatic system disorders) | 0 | 1 (2) | 0 | 2 (7)
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 | 1 (3) | 0 | 6 (28)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 (3)
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
Congenital, familial and genetic disorders - Other, difficulty concentrating (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 (1)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 1 (1)
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 (2)
Facial pain (General disorders) | 0 | 0 | 0 | 1 (1)
Fatigue (General disorders) | 0 | 1 (1) | 0 | 4 (6)
Fever (General disorders) | 0 | 0 | 0 | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 0 | 1 (1)
Flushing (Vascular disorders) | 0 | 0 | 0 | 2 (2)
Gastrointestinal disorders - Other, acid reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
General disorders and administration site conditions - Other, fluid retention (General disorders) | 0 | 0 | 0 | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
Headache (Nervous system disorders) | 0 | 0 | 0 | 3 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 1 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 2 (3) | 0 | 3 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 (2) | 0 | 3 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 (2) | 0 | 5 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 (2) | 0 | 5 (12)
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 (2)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
Localized edema (General disorders) | 0 | 0 | 0 | 1 (1)
Lymphocyte count decreased (Investigations) | 0 | 2 (6) | 0 | 6 (25)
Metabolism and nutrition disorders - Other, LDH elevated (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1)
Musculoskeletal and connective tissue disorder - Other, hand numbness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 (2)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
Neutrophil count decreased (Investigations) | 0 | 1 (1) | 0 | 2 (2)
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 (1)
Pain (General disorders) | 0 | 0 | 0 | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 4 (4)
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1)
Platelet count decreased (Investigations) | 0 | 0 | 0 | 4 (8)
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 3 (8)
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 (1)
Skin and subcutaneous tissue disorders - Other, peri-scapular pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 (3)
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
White blood cell decreased (Investigations) | 0 | 1 (3) | 0 | 4 (9)
General disorders and administration site conditions - Other (General disorders) | 0 | 0 | 0 | 1 (2) — Decreased breath sounds LLL
General disorders and administration site conditions - Other, oral thrush (General disorders) | 0 | 1 (1) | 0 | 1 (1)
General disorders and administration site conditions - Other, body aches (General disorders) | 0 | 0 | 0 | 1 (1)
General disorders and administration site conditions - Other, malaise (General disorders) | 0 | 1 (1) | 0 | 0
Musculoskeletal and connective tissue disorder - Other, jaw numbness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
Metabolism and nutrition disorders - Other, indigestion (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1)
Skin and subcutaneous tissue disorders - Other, rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form: Phase I portion consent (2014-12-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT01610570/ICF_000.pdf
  • Informed Consent Form: Phase II portion consent (2014-12-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT01610570/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT01610570/Prot_SAP_002.pdf